CLINICAL TRIAL: NCT06470425
Title: Optimizing Mental Health Management With AI-Guided (GenAIS TM) Dietary Supplementation: A Randomized Controlled Study
Brief Title: Optimizing Mental Health Management With AI-Guided (GenAIS TM) Dietary Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: S.LAB (SOLOWAYS) (Other)
Collaborators: Triangel Scientific (Industry); Center of New Medical Technologies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SW016
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-06

CONDITIONS: Mental Disorder
Keywords: AI-guided dietary supplementation; Genetic profiling; metabolic profiling; Depression management; anxiety management
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator)
  Interventions: Other: Standard therapy group
- AI-Guided Group (Experimental)
  Interventions: Other: AI-Guided group

INTERVENTIONS:
Other: Standard therapy group — Participants receive supplement prescriptions from a physician based on current standard practices, which include biochemical markers, genetic data, and metabolic profiles.
  Arms: Control Group
Other: AI-Guided group — Participants receive supplement prescriptions determined by GenAIS, is an AI system that considers genetic data, metabolic profiles, biochemical markers, and patient history.
  Arms: AI-Guided Group

SUMMARY:
The study "Optimizing Mental Health Management with AI-Guided (GenAIS TM) Dietary Supplementation" aimed to compare the effectiveness of AI-guided dietary supplement (DS) prescriptions versus standard physician-guided prescriptions in managing mental health disorders, specifically depression and anxiety. This 6-month randomized controlled trial included 160 participants diagnosed with major depressive disorder or generalized anxiety disorder. Participants were divided into two groups: one received DS based on physician judgment, and the other based on GenAIS AI system analysis. Primary outcomes focused on changes in mental health scores, while secondary outcomes included quality of life, metabolic markers, and DS adherence. Data collection involved genetic, metabolic, and clinical profiling, with ethical considerations ensuring participant confidentiality and informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years.
* Diagnosed with major depressive disorder (MDD) or generalized anxiety disorder (GAD) according to DSM-5 criteria.
* Moderate to severe symptoms as indicated by scores on HAM-D (≥17) for depression or GAD-7 (≥10) for anxiety.
* Stable on psychiatric medication for at least 3 months prior to the study.
* Willingness to provide genetic and metabolic data.
* Written informed consent.

Exclusion Criteria:

* Current or past history of severe psychiatric conditions such as schizophrenia, bipolar disorder, or other psychotic disorders.
* Current substance abuse or dependence within the last 6 months.
* Significant medical conditions like severe renal, hepatic, or cardiovascular diseases.
* Pregnancy or breastfeeding.
* Recent changes in psychiatric medication within the last 3 months.
* Participation in another clinical trial within the last 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the percent change in mental health scores (Hamilton Depression Rating Scale, Generalized Anxiety Disorder 7-item scale) for the AI-Guided group compared with the Control group. | 6 months
  The Hamilton Depression Rating Scale is a clinician-administered assessment used to measure the severity of depression in individuals. It consists of 17 to 21 items, with each item scored on a scale of 0 to 4 or 0 to 2.
  The Generalized Anxiety Disorder 7-item scale (GAD-7) is a self-administered questionnaire used to screen for and measure the severity of generalized anxiety disorder. It consists of 7 items, each scored from 0 (not at all) to 3 (nearly every day), with the total score ranging from 0 to 21. Higher scores indicate greater anxiety severity.

SECONDARY OUTCOMES:
Percent change in specific symptoms of depression and anxiety. | 6 months
Percent change in high-sensitivity C-reactive protein | 6 months
Percent change in body weight and body mass index | 6 months
Incidence of adverse effects related to dietary supplements. | 6 months
Number of Participant adherence to the prescribed dietary supplements regimen. | 6 months
Changes in quality of life score Short Form Health Survey | 6 months
  Short Form Health Survey, which has a score range from 0 to 100, to measure the quality of life in participants, with higher scores indicating better health and well-being
Changes in quality of life score World Health Organization Quality of Life | 6 months
  World Health Organization Quality of Life - BREF, which has a score range from 0 to 100, to measure the quality of life in participants, with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Center of New Medical Technologies, Novosibirsk, Novosibisk Region, Russia